CLINICAL TRIAL: NCT06221917
Title: Objective Assessment of Live-streaming Vs Face-to-face Teaching Method Effectiveness in Training Simple Wound Suturing Skill to Surgical Clerkship
Brief Title: Live-streaming Vs Face-to-face Teaching Method Effectiveness in Training Surgical Clerkship
Acronym: LS vs FTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelita Harapan University (Other)
Responsible Party: Principal Investigator, Freda Halim, Head of Surgery Department, Principal Investigator, Pelita Harapan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 011/K-LKJ/ETIK/I/2023
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Teaching Method
Keywords: Teaching method; Live-streaming; Face-to-face; Simple wound suturing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face (Active Comparator): Face-to-face teaching method
  Interventions: Other: Face-to-face
- Live-streaming (Experimental): Live-streaming teaching method
  Interventions: Other: Live-streaming

INTERVENTIONS:
Other: Face-to-face — FTF group are participants who will learn simple sutures physically present with the instructor in the same room.
  Arms: Face-to-face
Other: Live-streaming — One general surgeon (FH) will teach the participants how to do simple sutures on a mannequin, starting by explaining, then doing a live-demo step-by-step of simple wound suturing. The instructor uses a GoPro Hero 8 device on her head which is connected to the internet and produced live-streaming video, which will then be watched by LS group.
  Arms: Live-streaming

SUMMARY:
The goal of this observational study is to assess objectively whether teaching for simple wound sutures via Live-Streaming (LS) using Go-pro® has the same effectiveness as the traditional Face-to-face (FTF) teaching. The main question it aims to answer is whether training simple wound suturing skills to surgical clerkships via LS has the same effectiveness as the FTF training.

After initially doing pre-test, participants will be randomized into two groups: LS and FTF. After teaching exposure, the participants will be given 1 week period of self-training to master the skill (as such procedural skills require a period of self training before we examine the effect of teaching exposure). Afterwards, they underwent post-test again with the previously same examiner, using the same OSCE rubric to avoid bias. Researchers will compare if the LS and FTF groups to see if training simple wound suturing skills to surgical clerkships via LS has the same effectiveness as the FTF training.

ELIGIBILITY:
Inclusion Criteria:

* Surgery clerkships
* Willing to participate voluntarily and give consent to the study

Exclusion Criteria:

* Participants who drop out between 1 week period of pre-test and post-test
* Participants not willing to be involved in the teaching exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Post-test Scores | 1 week after teaching
  Post-test Objective Structured Clinical Exam (OSCE) scores Value ranges from 0 to 60. Higher score means better outcome, and vice versa.

SECONDARY OUTCOMES:
Numerical Differences of Pre-test and Post-test (Delta) | 1 week after teaching
  Numerical differences of Pre- and Post-Objective Structured Clinical Exam (OSCE) scores (Delta) Value ranges from -60 to 60. Higher numerical difference means better outcome, and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Freda Halim, Dr, dr, SpB, Principal Investigator — Pelita Harapan University
Locations (1):
- Pelita Harapan University, Tangerang, Banten, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made publicly available as part of an open access dataset.
Time Frame: The data will be available shortly after the study is finished, and will be available publicly for as long as needed.
Access Criteria: Open
URL: https://zenodo.org/

REFERENCES:
- [Background] Foo CC, Cheung B, Chu KM. A comparative study regarding distance learning and the conventional face-to-face approach conducted problem-based learning tutorial during the COVID-19 pandemic. BMC Med Educ. 2021 Mar 3;21(1):141. doi: 10.1186/s12909-021-02575-1. PMID 33658015
- [Background] McKechnie T, Levin M, Zhou K, Freedman B, Palter VN, Grantcharov TP. Virtual Surgical Training During COVID-19: Operating Room Simulation Platforms Accessible From Home. Ann Surg. 2020 Aug;272(2):e153-e154. doi: 10.1097/SLA.0000000000003999. No abstract available. PMID 32675522
- [Background] Doulias T, Gallo G, Rubio-Perez I, Breukink SO, Hahnloser D. Doing More with Less: Surgical Training in the COVID-19 Era. J Invest Surg. 2022 Jan;35(1):171-179. doi: 10.1080/08941939.2020.1824250. Epub 2020 Sep 22. PMID 32959688
- [Background] Navia A, Parada L, Urbina G, Vidal C, Morovic CG. Optimizing intraoral surgery video recording for residents' training during the COVID-19 pandemic: Comparison of 3 point of views using a GoPro. J Plast Reconstr Aesthet Surg. 2021 May;74(5):1101-1160. doi: 10.1016/j.bjps.2020.10.068. Epub 2020 Nov 8. No abstract available. PMID 33199220
- [Background] Song JSA, McGuire C, Vaculik M, Morzycki A, Plourde M. Cross sectional analysis of student-led surgical societies in fostering medical student interest in Canada. BMC Med Educ. 2019 Mar 8;19(1):77. doi: 10.1186/s12909-019-1502-5. PMID 30849966